CLINICAL TRIAL: NCT02959801
Title: Outcome of Percutaneous Mechanical Thrombectomy to Treat Acute Deep Venous Thrombosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12015C1038
Record Dates: First submitted 2016-07-19; First posted 2016-11-09 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Deep Venous Thrombosis
Keywords: Deep Venous Thrombosis; Percutaneous Mechanical Thrombectomy
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Percutaneous Mechanical Thrombectomy (Experimental): Percutaneous mechanical thrombectomy（PMT）uses a number of catheter-based mechanical devices to deliver the thrombolytic agent as well as to produce some combination of thrombus fragmentation, distribution of thrombolytic drugs throughout the thrombus, and/or thrombus aspiration.
  Interventions: Procedure: Percutaneous mechanical thrombectomy

INTERVENTIONS:
Procedure: Percutaneous mechanical thrombectomy — Aspirex catheters(Straub Medical AG, Wangs, Switzerland)

SUMMARY:
The purpose of this study was to compare the efficacy of Percutaneous mechanical thrombectomy (PMT) followed by standard anticoagulant therapy, with anticoagulation therapy alone, for the treatment of acute proximal lower extremity deep vein thrombosis.

DETAILED DESCRIPTION:
The conventional treatment of acute deep vein thrombosis (DVT) is anticoagulation therapy, as recommended in the international guidelines. Anticoagulation prevents recurrent venous thrombosis, pulmonary embolism, and death. Early thrombus removal is now considered as the standard of medical care for deep vein thrombosis (DVT). Early thrombus removal can offer the potential for early restoration of venous patency and preservation of valve function. Percutaneous mechanical thrombectomy (PMT) uses a number of catheter-based mechanical devices to deliver the thrombolytic agent as well as to produce some combination of thrombus fragmentation, distribution of thrombolytic drugs throughout the thrombus, and/or thrombus aspiration. The purpose of this study was to compare the efficacy of Percutaneous mechanical thrombectomy (PMT) followed by standard anticoagulant therapy, with anticoagulation therapy alone, for the treatment of acute proximal lower extremity deep vein thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* proven acute deep venous thrombosis, less than 21 days and who were referred to the interventional radiology department.

Exclusion Criteria:

* presence of subacute or chronic DVT more than 21 days in duration, inability to lie in the prone position required for intervention, terminal systemic disease requiring palliative treatment, active bleeding (from a gastric/duodenal ulcer or the cerebrovascular system), a haemorrhagic stroke within the previous year, an impaired bleeding-clotting profile, and any haemophilic disorder, or pregnancy.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
post-thrombotic syndrome | one year
  Clinical scoring was used to compare clinical symptoms and patient findings between the groups at six month and one year after treatment.

SECONDARY OUTCOMES:
complication | one year
  complication as death, bleeding, pulmonary embolism, recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tsinghua Chang Gung Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided